CLINICAL TRIAL: NCT02753543
Title: A Multi-center, Prospective, Single-arm, Open Label Phase II Study of Chidamide Combined With Chemotherapy in the Treatment of Peripheral T Cell Lymphoma
Brief Title: Chidamide Plus Chemotherapy in the Treatment of Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-PTCL-2016-01
Record Dates: First submitted 2016-04-19; First posted 2016-04-28 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chidamide plus previous chemotherapy (Experimental): Chidamide 20mg/d Biw p.o. on d1,4,8,11 for of each cycle for 3 cycles
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide

SUMMARY:
This is a single arm, prospective trial to evaluate the efficacy and safety of Chidamide in combination with previous chemotherapy in peripheral T cell lymphoma patients who did not achieve complete response after 3 cycles of chemotherapy in interim evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically verified peripheral T-cell lymphoma, partial response or stable disease after 3 cycles of CEOP (cyclophosphamide, epirubicin or doxorubicin, vincristine and prednisone) or CEOP(cyclophosphamide,vincristin,epirubicin and prednisone)/IVE (ifosfamide, epirubicin, etoposide)/GDP(Gemcitabine, Cis-platinum, Dexamethasone)
* Age ≧16 years, ≦75 years
* ECOG (Eastern Cooperative Oncology Group) =0,1,2
* No previous history of malignancy
* Radiologically measurable disease
* Life expectancy>6 months
* Informed consented

Exclusion Criteria:

* Active infectious disease requiring general antibiotics, anti-fungal or anti-virus therapy
* Lab at enrollment(unless caused by lymphoma)

  * Neutrophile<1.5*10^9/L
  * Platelet<75*10^9/L
  * Hemoglobulin<90g/L
  * ALT(alanine aminotransferase) or AST (aspartate aminotransferase ) >2*ULN,AKP(alkaline phosphatase) or bilirubin >1.5*ULN (upper limit of normal )
  * Creatinine>1.5*ULN
* Other uncontrollable medical condition that may that may interfere the participation of the study

  * Not able to comply to the protocol for mental or other unknown reasons
* Pregnant or lactation
* HIV infection

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
complete response | 21 days after 3 cycles of chidamide in combination with chemotherapy (each cycle is 21 days)

SECONDARY OUTCOMES:
Progression free survival | 1 year
Overall survival | 1 year
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Each cycle of treatment and then every 3 months for 1 year（each cycle is 21 days）

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No